CLINICAL TRIAL: NCT05848349
Title: Vitamin D Status, Its Determinants and IVF Outcomes Among Infertile Women in South-Western Sweden.
Brief Title: Vitamin D Status Among Infertile Women in Sweden
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Panagiotis Tsiartas, MD, PhD, Senior Consultant, M.D., Ph.D., Vastra Gotaland Region
Other Study IDs: VitDIVF
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Infertility, Female; Vitamin D Deficiency
MeSH Terms: conditions — Infertility, Female; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective cohort study is to learn about the overall and seasonal prevalence of vitamin D insufficiency and its determinants in a population of women with infertility who will go through in vitro fertilization in Sweden. The main questions it aims to answer are:

* What is the prevalence of vitamin D insufficiency?
* What are the determinants of this insufficiency? Participants will be asked to complete a questionnaire validated for dietary assessment of vitamin D intake and sun exposure habits and they will leave a blood sample for measurement of 25(OH)D concentration.

Researchers will compare the in vitro fertilization outcomes between women with vitamin D insufficiency and sufficiency to see if there is any difference.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-38 years, who will go through in vitro fertilization for infertility.

Exclusion Criteria:

* women who will go through pre-implantation genetic testing
* women who will go through sperm- or oocyte donation treatment
* Fertility preservation cycles

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women aged 18-38 who will go through in vitro fertilization during 2020-2021 (one year) for infertility at the Department of Obstetrics and Gynecology, Sahlgrenska University Hospital in Gothenburg, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of vitamin D insufficiency | September 2020 - August 2021
  Overall and seasonal prevalence of vitamin D insufficiency
Determinants of vitamin D insufficiency | September 2020 - August 2021
  Determinants (dietary, sun exposure habits) of vitamin D insufficiency

SECONDARY OUTCOMES:
In vitro fertilization outcomes | September 2020 - August 2021
  Pregnancy outcomes (biochemical pregnancy, clinical pregnancy, miscarriage, live birth) after in vitro fertilization between women with and without vitamin D insufficiency.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be made available on reasonable request.
Supporting Information: Study Protocol, SAP, ICF